CLINICAL TRIAL: NCT01230437
Title: The Effect of Montelukast on Inflammatory Responses of Nasal Epithelial Cells Cultured From Patients With Asthma, With and Without Concomitant Allergic Rhinitis
Brief Title: Montelukast and Nasal Epithelial Cell Inflammatory Responses in Asthma and Rhinitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr Garry Walsh, University of Aberdeen
Other Study IDs: MSD-36765-IISP; MT091 RGD 1265 (Other: University of Aberdeen)
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: montelukast; asthma; allergic rhinitis; nasal epithelial cells; inflammatory mediators
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- asthmatic patients taking montelukast: asthma with or without rhinitis

SUMMARY:
The airways of the lung are lined by specialised cells called airway epithelial cells. As well as being at the interface between the lungs and the air we breathe; airway epithelial cell (AEC) function is altered in people with respiratory diseases such as asthma. AEC secrete many mediators that contribute to asthma symptoms and these also contribute to asthmatic inflammation in the lungs. The study of such cells is difficult because of their location deep in the lungs. Nasal airway epithelial cells provide a useful and easily accessible model of model of lower airway cells. This study will examine whether the asthma medication Singulair (montelukast) can inhibit the inflammatory secretions of nasal AEC of asthmatic patents who also have allergic rhinitis compared with patients who have asthma alone. We will also examine if montelukast has differential modulating effects in these two patient groups.

DETAILED DESCRIPTION:
Hypothesis

The inflammatory secretory profile of nasal airway epithelial cells (NEC) cultured from asthmatics with concomitant allergic rhinitis (AR) will differ from that of NEC from patients with asthma alone. Treatment (in vitro and in vivo) with montelukast may have differential modulating effects in these two patient groups.

For the primary objective of this proposal we will use nasal AEC from asthmatics with or without concomitant AR as to ascertain differences in pro-inflammatory cytokine and chemokine production between these two groups and determine whether in vitro treatment with montelukast has a differential modulating effect on NEC secretion. In the secondary pilot study any modulating effects by montelukast on AEC secretion in vitro will be correlated with any in vivo response to montelukast withdrawal. This sub study will provide pilot data indicating whether in vivo response to montelukast can be predicted from in vitro effects on NEC.

ELIGIBILITY:
Inclusion Criteria:

* stable physician confirmed mild/moderate asthma (Steps 1-4 of BTS/SIGN guidelines <10 pack-year smoking histories Currently taking montelukast with a documented clinical history of benefit

Exclusion Criteria:

* Nasal corticosteroid therapy

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: For the primary study the investigators will identify 40 patients (aged 10-60) with with stable physician confirmed mild/moderate asthma (Steps 1-4 of BTS/SIGN guidelines [3]) with <10 pack-year smoking histories. Twenty of the subjects will have asthma and concomitant allergic rhinitis (asthma/AR) and 20 will have asthma alone.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Effect of montelukast on nasal epithelial cell secretion in vitro. | 12 months
  * Nasal AEC will be cultured from 20 patients with asthma and 20 patients with asthma and concomitant allergic rhinitis.
  * Unstimulated, TNFα (a surrogate for viral infection, a well known trigger of exacerbations) or allergen stimulated secretion of IL-6, IL-10, INFgamma TGFbeta, GM-CSF, eotaxin 1 & 2, RANTES and IL-8 by NEC will be measured. The in vitro inhibitory effects of a concentration range (10-6M to 10-10M) of montelukast will be assessed.

SECONDARY OUTCOMES:
Effect of 1-week montelukast withdrawal on clinical scores and pro-inflammatory cytokine output by nasal epithelial cells | 12 months
  * The secondary outcome of the study will be to examine the effect of withdrawal montelukast for 1-week on clinical scores and pro-inflammatory cytokine/ chemokine secretion by cultured NEC in montelukast-responsive patients with asthma (20 subjects) and asthma/AR (20 subjects).
  * The clinical scores and NEC secretory responses in these patients following montelukast withdrawal will be compared with the responses generated in the primary study i.e., while taking montelukast.

CONTACTS AND LOCATIONS:
Overall Officials: Garry M Walsh, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- [Background] McDougall CM, Blaylock MG, Douglas JG, Brooker RJ, Helms PJ, Walsh GM. Nasal epithelial cells as surrogates for bronchial epithelial cells in airway inflammation studies. Am J Respir Cell Mol Biol. 2008 Nov;39(5):560-8. doi: 10.1165/rcmb.2007-0325OC. Epub 2008 May 15. PMID 18483420